CLINICAL TRIAL: NCT06167772
Title: Effects of Leucine-enriched Branched-chain Amino Acid on Muscle Thickness, Interleukin-6, and Sequential Organ Failure Assessment Score in Critically Ill Patients
Brief Title: Leucine-enriched Branched-chain Amino Acid on Muscle Thickness, Interleukin-6, SOFA Score in Critical Illness
Acronym: SOFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Yohannessa Wulandari, M.Gizi, Sp GK, Principal Investigator, Clinical nutrition specialist; PhD student, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 23-09-1478
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Critical Illness; Muscle Wasting
Keywords: Leucine; Branched-chain amino acid; Muscle wasting; Critically-ill patients; Muscle thickness; Interleukin-6; Sequential organ failure assessment score
MeSH Terms: conditions — Critical Illness; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Branched-chain Amino Acid (BCAA) group (Experimental): branched-chain amino acid (bcaa) (ratio valine:leucine:isoleucine = 1.2:2:1) 40 g/day (leucine 19 g/day) form: powdered bcaa sealed in 8 g sachet package or bcaa parenteral 250 mL per bag.
  frequency: 1 sachet bcaa dissolved in oral nutrition supplement (standard nutrition) 5 times per day, or bcaa parenteral, or combination of bcaa enteral & parenteral.
  duration: 10 days standard nutrition: oral nutrition supplement (high protein) or parenteral with target energy of 20 kcal/kg BW/day standard neuromuscular electrical stimulation 30 minutes per day
  Interventions: Dietary Supplement: BCAA; Other: Standard nutrition; Other: Standard physiotherapy
- Control group (Placebo Comparator): No placebo. Not given intervention product. standard nutrition: oral nutrition supplement (high protein) or parenteral with target energy of 20 kcal/kg BW/day standard neuromuscular electrical stimulation 30 minutes per day
  Interventions: Other: Standard nutrition; Other: Standard physiotherapy

INTERVENTIONS:
Dietary Supplement: BCAA — branched-chain amino acid (bcaa) (ratio valine:leucine:isoleucine = 1.2:2:1) 40 g/day (leucine 19 g/day) form: powdered bcaa sealed in 8 g sachet package or bcaa parenteral 250 mL per bag.
  frequency: 1 sachet bcaa dissolved in oral nutrition supplement (standard nutrition) 5 times per day, or bcaa parenteral, or combination of bcaa enteral & parenteral.
  duration: 10 days
  Arms: Branched-chain Amino Acid (BCAA) group
Other: Standard nutrition — Target energy of 20 kcal/kg BW/day Target protein ratio protein:non-protein calorie 1:70
  Other Names: High protein oral nutritional supplementation
Other: Standard physiotherapy — A symmetric biphasic rectangular pulse was employed, with a frequency of 100 Hz, pulse width of 500 µs, Ton 5 s, Toff 25 s, ramp up of 1 s and ramp down of 1 s.
  Other Names: Neuromuscular electrical stimulation

SUMMARY:
The goal of this clinical trial study is to test effects of leucine-enriched branched-chain amino acid (BCAA) in critically ill patients. The main questions it aims to answer are: • How are the changes in muscle thickness between groups at baseline and end of study • Is there a decrease in interleukin-6 levels between groups at baseline and end of study • Is there a decrease in sequential organ failure assessment score between groups at baseline and end of study. Participants will be given leucine-enriched branched-chain amino acid 40 g/day enterally or parenterally for 10 days. Researchers will compare with control groups to see if there is any changes between groups at baseline and end of study.

DETAILED DESCRIPTION:
The goal of this clinical trial study is to test effects of leucine-enriched branched-chain amino acid (BCAA) in critically ill patients. The main questions it aims to answer are: • How are the changes in muscle thickness between groups at baseline and end of study • Is there a decrease in interleukin-6 levels between groups at baseline and end of study • Is there a decrease in sequential organ failure assessment score between groups at baseline and end of study. Participants will be given leucine-enriched branched-chain amino acid 40 g/day enterally or parenterally for 10 days. Researchers will compare with control groups to see if there is any changes between groups at baseline and end of study. Both groups will be given standard nutrition with target energy of 20 kcal/kg bodyweight(BW)/day and ratio of nitrogen:non-protein calorie 1:70 and neuromuscular electrical stimulation 30 minutes per day.

ELIGIBILITY:
Inclusion Criteria:

* new admission to intensive care unit (ICU) in first 24 hours
* aged 18-65 years
* SOFA score >= 4

Exclusion Criteria:

* pregnant
* ultrasound examination cannot be performed under these circumstances: deformities, open wounded, prosthetics on right leg, amputated above right patella
* body mass index <16 kg/m2
* chronic kidney disease stage 3-5
* diabetes mellitus uncontrolled blood glucose (BG) (BG >200 mg/dL)
* neuromuscular diseases with musculus quadriceps femoris dextra paralysis
* autoimmune diseases
* referral from another ICU

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Muscle thickness | 10 days
  Quadriceps femoris dextra muscle thickness between groups at baseline and end of study

SECONDARY OUTCOMES:
Interleukin-6 | 10 days
  Interleukin-6 levels between groups at baseline and end of study

OTHER OUTCOMES:
Sequential Organ Failure Assessment Score | 10 days
  Sequential Organ Failure Assessment Score between groups at baseline and end of study on scale 0-24

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region
  - Universitas Indonesia Hospital, Depok, West Java

REFERENCES:
- [Derived] Wulandari Y, Aditianingsih D, Sunardi D, Prasetyo M, Madjid AS, Nusdwinuringtyas N, Sutanto LB, Hardy G. High leucine branched-chain amino acids supplementation ameliorates quadriceps femoris muscle thickness reduction and attenuates interleukin-6 in critically ill patients: A randomised controlled trial. Clin Nutr ESPEN. 2025 Nov 29:102833. doi: 10.1016/j.clnesp.2025.11.153. Online ahead of print. PMID 41325937